CLINICAL TRIAL: NCT00055783
Title: A Phase II Study of Hu1D10 in Recurrent Hodgkin's Disease
Brief Title: Monoclonal Antibody Therapy in Treating Patients With Recurrent Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: SUMC-NCI-1951; CDR0000271198 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2003-03-06; First posted 2003-03-07 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2003-04

CONDITIONS: Lymphoma
Keywords: recurrent adult Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease | interventions — apolizumab

INTERVENTIONS:
Biological: apolizumab

SUMMARY:
RATIONALE: Monoclonal antibodies can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells.

PURPOSE: Phase II trial to study the effectiveness of monoclonal antibody therapy in treating patients who have progressive or recurrent Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate of patients with recurrent Hodgkin's lymphoma treated with monoclonal antibody Hu1D10.
* Determine the duration of response and progression-free survival of patients treated with this drug.
* Determine the toxicity of this drug in these patients.

OUTLINE: This is a multicenter study.

Patients receive monoclonal antibody Hu1D10 IV over 2 hours. Treatment repeats weekly for a total of 4 doses in the absence of disease progression or unacceptable toxicity.

Patients are followed at weeks 5 and 8 and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 9-24 patients will be accrued for this study within approximately 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed Hodgkin's lymphoma
* Progressive or recurrent disease after standard initial therapy
* At least 1 unidimensionally measurable lesion (at least 15 mm by conventional techniques)
* Patients in first relapse must be ineligible or unwilling to receive high-dose therapy and stem cell transplantation
* Evidence of Hu1D10 localization to Reed Sternberg cells by immunohistochemistry
* No known brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2 OR
* Karnofsky 60-100%

Life expectancy

* More than 6 months

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin normal
* AST and ALT no greater than 2.5 times upper limit of normal

Renal

* Creatinine normal OR
* Creatinine clearance at least 60 mL/min

Cardiovascular

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study participation
* HIV negative
* No known human anti-human antibody
* No prior allergic reaction to compounds of similar chemical or biological composition to monoclonal antibody Hu1D10
* No ongoing or active infection
* No other uncontrolled concurrent illness
* No psychiatric illness or social situation that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* See Chemotherapy

Chemotherapy

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* Prior second-line (or greater) high-dose therapy and stem cell transplantation allowed

Endocrine therapy

* Not specified

Radiotherapy

* At least 4 weeks since prior radiotherapy and recovered

Surgery

* Not specified

Other

* No other concurrent investigational agents
* No other concurrent anticancer agents or therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-07; Study Completion 2003-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra J. Horning, MD, Study Chair — Stanford University
Locations (1):
- Stanford University Medical Center, Stanford, California, United States